CLINICAL TRIAL: NCT05701813
Title: Effects of Inositols on Insulin Resistance in Children With Obesity (ONIRICO Trial)
Brief Title: The Study Aims to Investigate the Effects of Oral Inositols on Insulin-resistance in Children With Obesity.
Acronym: ONIRICO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Anita Morandi, Prof.ssa, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CESC 65739
Record Dates: First submitted 2023-01-19; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Prediabetic State; Dyslipidemias; Insulin Resistance
Keywords: INOSITOLS
MeSH Terms: conditions — Obesity; Prediabetic State; Dyslipidemias; Insulin Resistance | interventions — Cellulose

STUDY DESIGN:
Intervention Model Description: The children will be randomized into two arms, receiving either a mixture of inositols or placebo, for a period of 3 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation is performed by the nutraceutical supplier. Neither the participant, nor the investigator, nor the care provider, nor the outcome analyzer knows which arm the patient is assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INOSITOLS (Experimental): 4000 mg of myo-inositol and 300 mg of D-chiro-inositol. Once a day for 90 days.
  Interventions: Dietary Supplement: INOSITOLS
- PLACEBO (Placebo Comparator): Cellulose 4.3 grams once a day for 90 days.
  Interventions: Dietary Supplement: CELLULOSE

INTERVENTIONS:
Dietary Supplement: INOSITOLS — 4000 mg of myo-inositol and 300 mg of D-chiro-inositol. Once a day for 90 days.
  Arms: INOSITOLS
Dietary Supplement: CELLULOSE — 4.3 grams of cellulose once a day for 90 days.
  Arms: PLACEBO

SUMMARY:
The study aims to investigate the effects of oral inositols on insulin-resistance and metabolic variables (triglycerides, total cholesterol, HDL cholesterol) in children aged 8-12 years with obesity and insulin-resistance.

DETAILED DESCRIPTION:
Insulin-resistance is a condition, frequently related to obesity, that leads to cardio-metabolic complications in both children and adults, such as type 2 diabetes, hypertension, dyslipidemia and NAFLD. The best method to lower insulin-resistance is losing weight and doing physical activity, however changing lifestyle statistically reduces excess weight mildly. Also the genetic predisposition for a positive caloric balance, the difficulty in doing physical activity regularly and the metabolic and neuroendocrine responses aimed at preserving energy make it difficult to lose weight and/or improve one's insulin sensitivity. Infact, 80% of children chronicize their obesity into adulthood. For this reason, treatment should be based on both lifestyle changes and complementary approaches. Nutraceuticals can regulate physiological functions and are ideal candidates for children, since they are highly tolerated.

Myo-inositol and D-chiro-inositol are stereoisomers of sugar which, in combination with diacylglycerol (DAG), produce phosphatidylinositol (PI), precursor in the signalling of insulin and other hormones (growth factors and FSH). The insulin receptors leads to PI phosphorylation in PIP3, which activates kinases, such as Akt, that cause nuclear (cell proliferation) and cytoplasmatic (activation of glycogen synthetase) effetcs. It also activates phospholipase C, which hydrolyses PIP2 into DAG and IP3. IP3 leads to calcium liberation and moves GLUT4 to the surface of the cell membrane.

Inositols are also precursors of inositol-6 phosphate, which is important to promote adipocytes differentiation and fat oxidation.

Level A evidence shows that dietary supplements with one or both inositols used in women with PCOS to improve ovarian function, are highly effective also on insulin-sensitivity.

The aim of this study is to compare the efficacy of inositols versus placebo on insulin-resistance, measured with the HOMA-IR index, in a sample of children with obesity. As a secondary outcome, the study aims to enlight potential improvements in triglycerides, total cholesterol and HDL cholesterol.

This is a randomized, double-blind trial involving 56 children with obesity, aged 8 to 12 years, with insulin-resistance. The children will be randomized into two groups, receiving either a mixture of inositols or placebo, for a period of 3 months (90 days). During these 3 months, the children will be evaluated twice by dietitians (on day 45 and on day 90). Glucose, insulin and lipid profile will be assessed 0 to 30 days before the study beginning and at day 90 of the treatment period. During the visits, dietitians will take the anthropometric measurements, review the lifestyle goals and verify if the treatment is followed correctly (no more than one missed intake per week).

The mixture of inositols used contains 4000 mg of myo-inositol and 300 mg of D-chiro-inositol. The chosen dosages are based on two italian studies on young women with PCOS, where it's shown their effectiveness on matabolic risk factors and their high toerance. No dosage variation is required for the trial, since the weight of the evalueted children is similar to adults weight and there aren't differences in the clearance of the supplement. Side effects are rare (<1/1000) and mild (bloating, nausea and stomach ache).

The difference in the pre-post treatment HOMA-IR and lipids changes between the two arms will be analyzed with the Student t Test for independent samples, presuming a gaussian distribution of the variable changes. The expected change difference between arms considered clinically significant and used to calculate the arm size is at least 1 standard deviation. The supplement will be considered tollerable if the frequency of side effects will be not significantly different between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Age under 12 and over 8 years
* Presence of obesity defined by BMI > 95th percentile of BMI based on the growth curves of the Italian Society of Pediatric Endocrinology and Diabetology (Cacciari curves)
* Presence of HOMA-IR value (insulin x glycaemia/22.5: marker of insulin resistance) > 75th percentile of a reference pediatric population from Verona

Exclusion Criteria:

* Diabetes mellitus
* Current chronic disease with systemic inflammation
* Use of drugs acting on insulin sensitivity (e.g. steroids)
* Use of food or vitamin supplements up to one month before blood sampling
* Puberty in progress

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy on insulin-resistance, measured with the HOMA-IR index | 90 days
  Difference in HOMA-IR index change across arms

SECONDARY OUTCOMES:
Improvements in triglycerides, total cholesterol and HDL cholesterol. | 90 days
  Difference in changes of metabolic variables over time across arms

OTHER OUTCOMES:
Effect on BMI (Body Mass Index) | 90 days
  Difference in the change of BMI over time across arms

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chatree S, Thongmaen N, Tantivejkul K, Sitticharoon C, Vucenik I. Role of Inositols and Inositol Phosphates in Energy Metabolism. Molecules. 2020 Nov 1;25(21):5079. doi: 10.3390/molecules25215079. PMID 33139672
- [Background] Shokrpour M, Foroozanfard F, Afshar Ebrahimi F, Vahedpoor Z, Aghadavod E, Ghaderi A, Asemi Z. Comparison of myo-inositol and metformin on glycemic control, lipid profiles, and gene expression related to insulin and lipid metabolism in women with polycystic ovary syndrome: a randomized controlled clinical trial. Gynecol Endocrinol. 2019 May;35(5):406-411. doi: 10.1080/09513590.2018.1540570. Epub 2019 Jan 4. PMID 30608001
- [Background] Fruzzetti F, Perini D, Russo M, Bucci F, Gadducci A. Comparison of two insulin sensitizers, metformin and myo-inositol, in women with polycystic ovary syndrome (PCOS). Gynecol Endocrinol. 2017 Jan;33(1):39-42. doi: 10.1080/09513590.2016.1236078. Epub 2016 Nov 3. PMID 27808588
- [Background] Pizzo A, Lagana AS, Barbaro L. Comparison between effects of myo-inositol and D-chiro-inositol on ovarian function and metabolic factors in women with PCOS. Gynecol Endocrinol. 2014 Mar;30(3):205-8. doi: 10.3109/09513590.2013.860120. Epub 2013 Dec 19. PMID 24351072
- [Background] Kachhawa G, Senthil Kumar KV, Kulshrestha V, Khadgawat R, Mahey R, Bhatla N. Efficacy of myo-inositol and d-chiro-inositol combination on menstrual cycle regulation and improving insulin resistance in young women with polycystic ovary syndrome: A randomized open-label study. Int J Gynaecol Obstet. 2022 Aug;158(2):278-284. doi: 10.1002/ijgo.13971. Epub 2021 Nov 10. PMID 34624138
- [Background] Bahadur A, Arora H, Ravi AK, Naithani M, Bahurupi Y, Chaturvedi J, Ajmani M, Mundhra R. Comparison of Clinical, Metabolic and Hormonal Effects of Metformin Versus Combined Therapy of Metformin With Myoinositol Plus D-Chiro-Inositol in Women With Polycystic Ovary Syndrome (PCOS): A Randomized Controlled Trial. Cureus. 2021 Jun 7;13(6):e15510. doi: 10.7759/cureus.15510. eCollection 2021 Jun. PMID 34268040
- [Background] Maffeis C, Morandi A. Body composition and insulin resistance in children. Eur J Clin Nutr. 2018 Sep;72(9):1239-1245. doi: 10.1038/s41430-018-0239-2. Epub 2018 Sep 5. PMID 30185840
- [Background] Rajjo T, Mohammed K, Alsawas M, Ahmed AT, Farah W, Asi N, Almasri J, Prokop LJ, Murad MH. Treatment of Pediatric Obesity: An Umbrella Systematic Review. J Clin Endocrinol Metab. 2017 Mar 1;102(3):763-775. doi: 10.1210/jc.2016-2574. PMID 28359101
- [Background] Hayes AJ, Carrello JP, Kelly PJ, Killedar A, Baur LA. Looking backwards and forwards: tracking and persistence of weight status between early childhood and adolescence. Int J Obes (Lond). 2021 Apr;45(4):870-878. doi: 10.1038/s41366-021-00751-3. Epub 2021 Feb 8. PMID 33558641
- [Background] Elks CE, den Hoed M, Zhao JH, Sharp SJ, Wareham NJ, Loos RJ, Ong KK. Variability in the heritability of body mass index: a systematic review and meta-regression. Front Endocrinol (Lausanne). 2012 Feb 28;3:29. doi: 10.3389/fendo.2012.00029. eCollection 2012. PMID 22645519
- [Background] Llewellyn C, Wardle J. Behavioral susceptibility to obesity: Gene-environment interplay in the development of weight. Physiol Behav. 2015 Dec 1;152(Pt B):494-501. doi: 10.1016/j.physbeh.2015.07.006. Epub 2015 Jul 10. PMID 26166156
- [Background] Silventoinen K, Jelenkovic A, Sund R, Yokoyama Y, Hur YM, Cozen W, Hwang AE, Mack TM, Honda C, Inui F, Iwatani Y, Watanabe M, Tomizawa R, Pietilainen KH, Rissanen A, Siribaddana SH, Hotopf M, Sumathipala A, Rijsdijk F, Tan Q, Zhang D, Pang Z, Piirtola M, Aaltonen S, Oncel SY, Aliev F, Rebato E, Hjelmborg JB, Christensen K, Skytthe A, Kyvik KO, Silberg JL, Eaves LJ, Cutler TL, Ordonana JR, Sanchez-Romera JF, Colodro-Conde L, Song YM, Yang S, Lee K, Franz CE, Kremen WS, Lyons MJ, Busjahn A, Nelson TL, Whitfield KE, Kandler C, Jang KL, Gatz M, Butler DA, Stazi MA, Fagnani C, D'Ippolito C, Duncan GE, Buchwald D, Martin NG, Medland SE, Montgomery GW, Jeong HU, Swan GE, Krasnow R, Magnusson PK, Pedersen NL, Dahl Aslan AK, McAdams TA, Eley TC, Gregory AM, Tynelius P, Baker LA, Tuvblad C, Bayasgalan G, Narandalai D, Spector TD, Mangino M, Lachance G, Burt SA, Klump KL, Harris JR, Brandt I, Nilsen TS, Krueger RF, McGue M, Pahlen S, Corley RP, Huibregtse BM, Bartels M, van Beijsterveldt CE, Willemsen G, Goldberg JH, Rasmussen F, Tarnoki AD, Tarnoki DL, Derom CA, Vlietinck RF, Loos RJ, Hopper JL, Sung J, Maes HH, Turkheimer E, Boomsma DI, Sorensen TI, Kaprio J. Differences in genetic and environmental variation in adult BMI by sex, age, time period, and region: an individual-based pooled analysis of 40 twin cohorts. Am J Clin Nutr. 2017 Aug;106(2):457-466. doi: 10.3945/ajcn.117.153643. Epub 2017 Jul 5. PMID 28679550
- [Background] Roth CL, Melhorn SJ, De Leon MRB, Rowland MG, Elfers CT, Huang A, Saelens BE, Schur EA. Impaired Brain Satiety Responses After Weight Loss in Children With Obesity. J Clin Endocrinol Metab. 2022 Jul 14;107(8):2254-2266. doi: 10.1210/clinem/dgac299. PMID 35544121
- [Background] Fernandez I, Canet O, Gine-Garriga M. Assessment of physical activity levels, fitness and perceived barriers to physical activity practice in adolescents: cross-sectional study. Eur J Pediatr. 2017 Jan;176(1):57-65. doi: 10.1007/s00431-016-2809-4. Epub 2016 Nov 17. PMID 27858223
- [Background] Cacciari E, Milani S, Balsamo A, Spada E, Bona G, Cavallo L, Cerutti F, Gargantini L, Greggio N, Tonini G, Cicognani A. Italian cross-sectional growth charts for height, weight and BMI (2 to 20 yr). J Endocrinol Invest. 2006 Jul-Aug;29(7):581-93. doi: 10.1007/BF03344156. PMID 16957405
- [Background] Takemoto K, Deckelbaum RJ, Saito I, Likitmaskul S, Morandi A, Pinelli L, Ishii E, Kida K, Abdalla M. Adiponectin/resistin levels and insulin resistance in children: a four country comparison study. Int J Pediatr Endocrinol. 2015;2015(1):2. doi: 10.1186/1687-9856-2015-2. Epub 2015 Jan 15. PMID 25904939
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714